CLINICAL TRIAL: NCT02118402
Title: In Home Iron Fortification in Kenyan Infants: Effect of Co-supplementation With Galactooligosaccharides (GOS) on the Gut Microbiota Composition and the Effectiveness of Iron Supplementation
Brief Title: Iron and Prebiotics Fortification in Kenyan Infants
Acronym: Iro'n'Pre
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DSM-2-70790-11
Record Dates: First submitted 2014-04-10; First posted 2014-04-21 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Anemia; Iron Deficiency; Diarrhea; Malaria; Respiratory Tract Infections (RTI); Antibiotics; Gut Inflammation; Prebiotics; Vaccine Response
MeSH Terms: conditions — Anemia; Iron Deficiencies; Diarrhea; Malaria; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fortified maize porridge (MNP) (Active Comparator): The MNP contains 400 µg Vitamin A, 5 µg Vitamin D, 5 mg Tocopherol Equivalent, 0.5 mg Thiamine, 0.5 mg Riboflavin, 0.5 mg Vitamin B6 , 90 µg Folic Acid, 6 mg Niacin, 0.9 µg Vitamin B12, 30 mg Vitamin C, 0.56 mg Copper, 90 µg Iodine, 17 µg Selenium, 4.1 mg Zinc, 190 Phytase-units, maltodextrin carrier (added up to 11g)
  Interventions: Dietary Supplement: Fortified maize porridge
- Fortified maize porridge (MNP+Fe) (Active Comparator): The MNP contains 400 µg Vitamin A, 5 µg Vitamin D, 5 mg Tocopherol Equivalent, 0.5 mg Thiamine, 0.5 mg Riboflavin, 0.5 mg Vitamin B6 , 90 µg Folic Acid, 6 mg Niacin, 0.9 µg Vitamin B12, 30 mg Vitamin C, 0.56 mg Copper, 90 µg Iodine, 17 µg Selenium, 4.1 mg Zinc, 190 Phytase-units, plus 2.5 mg Fe as ferrous fumarate and 2.5 mg Fe as NaFeEDTA, maltodextrin carrier (added up to 11g)
  Interventions: Dietary Supplement: Fortified maize porridge
- Fortified maize porridge (MNP+Fe+GOS) (Active Comparator): The MNP contains 400 µg Vitamin A, 5 µg Vitamin D, 5 mg Tocopherol Equivalent, 0.5 mg Thiamine, 0.5 mg Riboflavin, 0.5 mg Vitamin B6 , 90 µg Folic Acid, 6 mg Niacin, 0.9 µg Vitamin B12, 30 mg Vitamin C, 0.56 mg Copper, 90 µg Iodine, 17 µg Selenium, 4.1 mg Zinc, 190 Phytase-units, 2.5 mg Fe as ferrous fumarate and 2.5 mg Fe as NaFeEDTA plus 7.5 g of galactooligosaccharides given as 10.5 g GOS-75, maltodextrin carrier (added up to 11g)
  Interventions: Dietary Supplement: Fortified maize porridge

INTERVENTIONS:
Dietary Supplement: Fortified maize porridge — Maize porridge will be home-fortified with either A) MNP, B) MNP+Fe, C) MNP+Fe+GOS

SUMMARY:
Iron deficiency and anemia are health issues affecting mainly infants and women in developing countries. Iron deficiency in infancy can have long-lasting impact on cognitive and motor development of the child. Iron fortification has shown to be effective against anemia. However, in areas with a high burden of infectious diseases iron may increase the risk of unfavorable gut microbiota composition possibly influencing diarrhea prevalence. Therefore we want to assess the effects of home fortification of complementary food with two iron-containing micronutrient powders (MNPs) with and without the addition of a prebiotic (7.5 g of galactooligosaccharides as GOS-75) compared to a control on the composition of the gut microbiota of Kenyan infants. In addition, iron deficiency may iimpair adaptive immunity. Following Kenyan Minstry of Health guidelines, infants receive their first measles vaccine at 9 months. In this study we will use an MNP with a moderate iron dose of 5 mg, with 2.5 mg of Fe as NaFeEDTA and 2.5 mg of Fe as ferrous fumarate (+Fe). There will be 3 study groups MNP, MNP+Fe and MNP+Fe+GOS. The infants will be enrolled in the study at the age of 6-10 months and will consume a home-fortified maize porridge for four months. At baseline and endpoint (after 4 months of intervention), we will collect blood samples of the infants in order to assess anemia, iron status, and inflammation. In addition, we will assess the effect of iron supplementation on measles vaccine response. Fecal samples (from child and mother) will be collected at baseline, 3 weeks and at endpoint in order to evaluate the changes in gut microbiota and gut inflammation.

During the intervention, in a sub-group of children who receive broad-spectrum antibiotics, we will compare how the three different interventions modify the effect of antibiotics on the infant gut microbiota. We will opportunistically select children that are enrolled in the study and who become ill, and who are prescribed antibiotics by the local health care team, according to the local standard of care in the study area. Five additional stool samples from these children will be collected (day 0 (before the first antibiotic dose), 5, 10, 20 and 40) to evaluate the changes in the gut microbiota and gut inflammation.

Three years after the study end, we would like to collect a blood and stool sample from the children and examine the iron status and gut microbiome respectively.

DETAILED DESCRIPTION:
Fifty infants per group will be enrolled (n=150) and randomly divided in three groups, from those identified in selected villages in the catchment area of the Kikoneni Health Clinic in southern coastal Kenya, about 2 hours south of Mombasa. All children whose caregivers agree to participate in the study will have their iron status assessed by measurement of hemoglobin (Hb), erythrocyte zinc protoporphyrin (ZPP), serum ferritin (SF) and serum transferrin receptor (TfR). Enrolled subjects will be randomized into three groups. Group 1 will receive the MNP alone, group 2 will receive an identical MNP with iron (2.5 mg Fe as NaFeEDTA and 2.5 mg as ferrous fumarate), and group 3 will receive the MNP with iron (2.5 mg Fe as NaFeEDTA and 2.5 mg as ferrous fumarate) and 7.5 mg of galactooligosaccharides as GOS-75. Each household will receive 2 kg of maize meal per week and the caregivers of the participating children will be shown how to prepare a maize porridge, which is the most widely-used local complementary food. This maize meal will be provided free-of-charge to all participating families. The caregiver will add one MNP sachet each day to a portion of maize porridge, and feed the entire portion to the infant. The Kikoneni Clinic will serve as the collection point for the MNPs, the monitoring center for surveillance of infant health, as well as the blood and stool collection point.

At baseline and at endpoint of the intervention (after 4 months), a blood sample will be collected from the infants for measurement of Hb, SF, TfR and ZPP to define anemia and iron status and C-reactive protein (CRP) to define systemic inflammation status. In addition, anti-measles Serum IgG will be measured, as infants receive their first measles vaccination at 9 months, following Kenyan Ministry of Health guidelines. At baseline, after 3 weeks and after 4 month, a stool sample will be collected from both the infant and his/her mother, for measurement of the gut microbiota and gut inflammation.The mothers will be trained to collect the stool samples at home in a provided container with a tight, screw-top lid, that includes an Anerocult® sachet to create an anaerobic environment. At these 3 timepoints (baseline, after 3 weeks and after 4 month) the mother will bring in the two stool samples of the same day, where they will be labeled and kept at 4°C. The samples will be then transferred to the central lab, filled in 2 ml Eppendorf tubes, labelled and frozen at -20°C.

In addition, compliance and morbidity will be assessed weekly during the distribution of the MNPs. The children will be checked and referred to the health center clinicians whenever indicated by the clinical history. In the case of fever, a rapid malaria test (RTD) kit will be performed according to local guidelines. If the test results positive, the child will be treated for presumptive malaria, mild malaria cases will be treated at Kikoneni clinic as per WHO Integrated management of childhood illness (IMCI) guidelines. Cases of diarrhea will be treated according to the local standard of care including oral rehydration salt and, if necessary, antibiotics. If deemed necessary by the Kikoneni clinical management, the study team will support the clinic in re stocking ORS, iron supplements and antimalaric drugs for the study duration.

Anthropometry (weight, height, age and sex) will be recorded at baseline and endpoint using standardized procedures to calculate the prevalence of child stunting. The measurements will be done twice and the average used for data analysis. The data analysis software WHO Anthro (WHO, Geneva Switzerland) will be used to calculate the prevalence of stunting among this infant population.

To investigate the effect of oral antibiotics on the infant gut microbiota we will select the first 12 infants of each of the three study groups that become ill during the study and receive broad-spectrum antibiotic treatment. We will also select 6 non-treated controls from each study group matched for sex and weeks of MNP consumption. A total of n=54 children will be included in this sub study and we will collect five additional stool samples from the selected children to determine the gut microbiota composition. The first stool sample will be collected before starting the antibiotic treatment (day 0). Thereafter, a stool sample will be collected at day 5, 10, 20 and 40. Stool samples will be collected as described above. Besides these additional stool samples the children continue the intervention according to the main protocol.

A breast milk sample will be collected from 90 mothers at two time points (week 3 and week 16). These samples will be analyzed for the concentration of human milk oligosaccharides, a potential source of natural prebiotics.

Three years after the end of the study, we would like to examine iron status and gut microbiota of these children and determine whether the differences observed after the intervention persist or if they all converge and have a similar microbiome profile. In addition, we will measure anti-measles serum IgG, as infants received their second measles vaccine at 18 months following Kenyan Ministry of Health guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age of 6-10 months at baseline
* Assessment of good health as assessed by professional staff at Kikoneni Health Clinic.
* Willingness of their caregiver to provide informed consent

Exclusion Criteria:

* Hemoglobin <7g/dL; these participants will be referred for treatment at the local health clinic according to the guidelines of Kenya Ministry of Health.
* Participants taking part in other studies requiring the drawing of blood.
* Chronic or acute illness or other conditions that in the opinion of the PI or co-researchers would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol.
* Not planning long-term residence in study site
* Participants who are taking iron-containing food supplements or tablets/drops.

Ages: 6 Months to 14 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 155 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The co-primary outcomes are the gut microbiome and gut inflammation | Change from baseline to 3 weeks and 16 weeks
  We will measure key commensal and pathogenic members of the fecal gut microbiota of the infants using qPCR and 16S rDNA sequencing. We will measure fecal calprotectin and serum intestinal fatty acid binding protein as markers of gut inflammation and enterocyte injury. The changes in these measurements during the intervention will be compared among the three groups.

SECONDARY OUTCOMES:
Iron status and systemic inflammation | Change from baseline to endpoint (16 weeks)
  We will assess serum ferritin, soluble transferrin receptor, erythrocyte zinc protoporphyrin and hemoglobin to define the iron status. C-reactive protein to assess systemic inflammatory status. The changes in these measurements during the intervention will be compared among the three groups.
Anthropometry | Change from baseline to endpoint (16 weeks)
  Anthropometric data (weight, height, age and sex) will be recorded using standardized procedures to calculate the prevalence of child stunting. Measurements will be conducted at the start of the intervention and after 4 months (end point). The data analysis software WHO Anthro (WHO, Geneva Switzerland) will be used to calculate the prevalence of stunting among this infant population. The changes in these measurements during the intervention will be compared among the three groups.
Child to -mother transmission of gut microbiota | Change from baseline to 3 weeks and endpoint (16 weeks)
  We will measure key commensal and pathogenic members of the fecal gut microbiota of the mothers using qPCR and pyrosequencing. We will measure fecal calprotectin and serum and fecal zonulin as markers of gut inflammation. The changes in these measurements during the intervention will be compared among the three groups of mothers, and correlations will be done to assess associations of the variables within the mother-child pairs.
Gut microbiota and gut inflammation during and after an oral antibiotic treatment | Change from baseline day 0 (prior to antibiotic administration) to day 5, 10, 20 and 40
  We will measure key commensal and pathogenic members of the fecal gut microbiota of the infants using qPCR and pyrosequencing. We will measure fecal calprotectin and serum and fecal zonulin as markers of gut inflammation. The changes in these measurements during and after an oral antibiotic treatment will be assessed and compared between the three groups.
Morbidity | Weekly assessment from baseline to endpoint (16 weeks)
  Morbidity data (fever, cough, diarrhea, bloody and mucous stool) will be assessed weekly with a questionnaire. The frequency of these morbidities during the intervention will be compared among the three groups.

OTHER OUTCOMES:
Human milk oligosaccharides in breast milk | Sampling time points at week 3 and week 16
  Breast milk from n=90 mothers will be analyzed to quantify human milk oligosaccharides concentration.
Long term gut microbiota composition | Change from endpoint to 3 years after study end
  We will measure key commensal and pathogenic members of the fecal gut microbiota of the infants using qPCR and pyrosequencing. We will measure fecal calprotectin and fecal zonulin as markers of gut inflammation. The changes in these measurements compared to endpoint will be assessed and compared between the three intervention groups
Long term iron status and systemic inflammation | Change from endpoint to 3 years after study end
  We will assess serum ferritin, soluble transferrin receptor and hemoglobin to define the iron status. Using C-reactive protein and alpha-1-acid glycoprotein we will assess inflammatory status. The changes in these measurements during the intervention will be compared among the three groups.
Primary vaccine response | anti-measels serum IgG and avidity at age 12months (endpoint intervention)
  We will determine anti-measles serum IgG and IgG avidity to assess vaccine response
Secondary vaccine response | anti-measels serum IgG and avidity at 3 years after study end
  We will determine anti-measles serum IgG and IgG avidity to assess vaccine response

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zimmermann, MD, Principal Investigator — ETH Zurich
Locations (1):
- Kikoneni Health Center, Kikoneni, Kwale County, Kenya

REFERENCES:
- [Derived] Paganini D, Uyoga MA, Kortman GAM, Cercamondi CI, Winkler HC, Boekhorst J, Moretti D, Lacroix C, Karanja S, Zimmermann MB. Iron-containing micronutrient powders modify the effect of oral antibiotics on the infant gut microbiome and increase post-antibiotic diarrhoea risk: a controlled study in Kenya. Gut. 2019 Apr;68(4):645-653. doi: 10.1136/gutjnl-2018-317399. Epub 2018 Nov 17. PMID 30448776
- [Derived] Paganini D, Uyoga MA, Kortman GAM, Cercamondi CI, Moretti D, Barth-Jaeggi T, Schwab C, Boekhorst J, Timmerman HM, Lacroix C, Karanja S, Zimmermann MB. Prebiotic galacto-oligosaccharides mitigate the adverse effects of iron fortification on the gut microbiome: a randomised controlled study in Kenyan infants. Gut. 2017 Nov;66(11):1956-1967. doi: 10.1136/gutjnl-2017-314418. Epub 2017 Aug 3. PMID 28774885